CLINICAL TRIAL: NCT04081714
Title: Intermediate Expanded Access Protocol With CNM-Au8 for Multiple Sclerosis
Brief Title: Intermediate Expanded Access Protocol CNMAu8.EAP03
Status: Temporarily not available | Type: Expanded Access
Sponsor: Clene Nanomedicine (Industry)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Sponsor
Other Study IDs: CNMAu8.EAP03
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: MS; Gold; Nanoparticle; Expanded access; Au8; CNMAu8
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: CNM-Au8 — CNM-Au8 is an aqueous suspension of clean surfaced faceted nanocrystals consisting of gold atoms self-organized into crystals of various geometrical shapes (hexagonal bi-pyramid, pentagonal bipyramid, tetrahedron, decahedron, planar spheroids). Highly pure elemental Au nanocrystals are suspended in USP purified deionized water buffered with 0.546 mg/mL (6.5 mM) sodium bicarbonate (NaHCO3) nominally concentrated to 0.5 mg/L (500 ppm). CNM-Au8 will be administered orally in volumes of 60 mL from single-dose HDPE containers. Participants will orally receive 30 mg of CNM-Au8 once daily.
  Other Names: Nanocrystalline gold

SUMMARY:
This is a single-center intermediate expanded access program to provide access to the investigational product, CNM-Au8, up to 25 participants diagnosed with Multiple Sclerosis.

DETAILED DESCRIPTION:
This is an intermediate expanded access program to provide access to the investigational product, CNM-Au8, for up to 25 participants. All participants will receive open label treatment with CNM-Au8 30 mg orally.

The safety and efficacy of CNM-Au8 treatment in MS participants will be evaluated. Scheduled visits will occur at the baseline visit, week 6 visit, week 12, and then every 12-weeks thereafter at the participating clinic(s). Optional remote data collection via telemedicine and/or home healthcare visits are permitted commencing with the week 12 visit. Clinical safety laboratory monitoring including urinalysis, a chemistry panel (e.g., CMP) and a hematology panel (e.g., CBC) will be conducted at the screening/baseline visit and at each scheduled visit incorporating safety laboratory assessments.

Participants who meet the inclusion criteria and none of the exclusionary criteria may be enrolled into the EAP.

The program and participant visits will continue for a total of 96-weeks of treatment. Four weeks following treatment discontinuation, a safety follow-up visit will be conducted.

Investigational product may be shipped by the site to participants who do not attend an in-clinic visit.

The EAP may be discontinued at the Sponsor's sole discretion if: (i) there is insufficient funding to maintain the EAP, (ii) the Sponsor is unable to produce sufficient supply of the investigational product to meet clinical trial obligations, (iii) CNM-Au8 receives marketing authorization within the United States, or (iv) continued support of the EAP risks further clinical development of CNM-Au8.

ELIGIBILITY:
Participants in the EAP must meet all the following inclusion criteria:

1. Able to understand and give written informed consent.
2. Male or female participants aged 18 years or greater (inclusive) at the time of informed consent.
3. Participants with a neurologist confirmed diagnosis of MS per the 2017 McDonald criteria of relapsing MS (RMS), non-active secondary progressive MS (NA-SPMS), or primary progressive MS (PPMS).
4. Participant can consume up to 120 mL of the investigational drug suspension daily.
5. Participant is not adequately treated by current standard of care DMT, which is evidenced by: progression independent of relapse activity (PIRA) based on an EDSS change of 0.5 or more over a 6-month period where the initial EDSS was 4.0 or more, OR an EDSS increase of 1.0 or more if over a 6-month period where the initial EDSS was 2.0 or more, AND the participant has been treated with an MS immunomodulatory disease modifying treatment (DMT) including S1P drugs (e.g., fingolimod, ponesimod, ozanimod), natalizumab, cladribine, a B-cell depleting therapy (e.g., ocrelizumab, ofatumumab), or other appropriate DMTs for at least the prior 6-months, OR has demonstrated an EDSS increase per the criteria above despite at least a 6-month period of prior immunomodulatory DMT treatment that was subsequently discontinued due lack of response or intolerance to treatment.
6. Participant has an EDSS score of greater than or equal to 2.0 and less than or equal to 6.5.

Participants may not be enrolled if they meet any of the following exclusion criteria:

1. A clinical relapse within the prior six months. NA-SPMS and PPMS participants may not have had a history of gadolinium enhancing lesions within the prior 24-months.
2. History of significant major medical condition(s) that may interfere with the conduct of the EAP or interpretation of the EAP results as determined by the Investigator.
3. Based on the Investigator's judgment, participants who may have difficulty complying with the protocol and/or study procedures.
4. History of any clinically significant abnormality in hematology, blood chemistry, ECG, or physical examination not resolved by the Screening/Baseline visit.
5. Participant has clinically significant findings at the Screening/Baseline visit on standard hepatic, hematologic, or renal safety assays, including but not limited to: (i) ALT or AST ≥ 3 times upper limits of normal, (ii) direct (conjugated) with bilirubin ≥2 times upper limits of normal, (iii) Child-Pugh Classification B (moderate) or C (severe), (iv) low platelet counts (< 150 x 109 per liter), (v) eosinophilia (absolute eosinophil count of ≥ 500 eosinophils per microliter), (vi) serum creatinine >1.2 mg/dL, or (vii) eGFR < 45 ml/min per 1.73 m2.
6. Females who are pregnant, have a positive pregnancy test, are nursing, or who plan to get pregnant during participation in the EAP or within 6 months of the ending participation in the EAP.
7. Women of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control during the study and for 6 months following completion of study participation.
8. Participants with a history of gold allergy.
9. Participant is considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating any active or intermittent suicidal ideation.
10. Participants with a history of any of the following: a. History of human immunodeficiency virus (HIV), hepatitis C (HepC) virus antibody, or hepatitis B (HepB) virus antibody without history of previous HepB vaccination. b. History or evidence of substance abuse or alcohol abuse within 5- years prior to Screening, including alcoholism; or severe tobacco use (>1 pack/day). c. Any history of previous malignancy, with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix, post documented full resections, with clean margins.
11. Current treatment with immunosuppressive or immunomodulatory therapy other than those approved for the treatment of MS.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States